CLINICAL TRIAL: NCT05479149
Title: Effectiveness of a Novel Device for Cervical Training in Cervicogenic Headache. Randomized Clinical Trial.
Brief Title: Effectiveness of a Novel Device for Cervical Training in Cervicogenic Headache.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universitat Internacional de Catalunya (Other)
Responsible Party: Principal Investigator, Pilar Pardos Aguilella, Colaborator Lecturer in Physiotherapy, Universitat Internacional de Catalunya
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: C.P-C.I.PI21/357
Record Dates: First submitted 2022-07-25; First posted 2022-07-29 (Actual); Last update posted 2023-01-27 (Actual); Status verified 2023-01

CONDITIONS: Cervicogenic Headache
Keywords: neck muscles; headache pain; muscle weakness; telerehabilitation; exercise therapy
MeSH Terms: conditions — Post-Traumatic Headache; Muscle Weakness | interventions — Therapeutics

STUDY DESIGN:
Intervention Model Description: This will be a randomized controlled trial with 2 different groups
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental: Training protocol with the cervical device for treatment (CDAT). (Experimental): Endurance training program of deep cervical flexors and deep cervical extensors with the cervical device for treatment.
  Interventions: Other: Training protocol with the cervical device for treatment (CDAT).
- Conventional training protocol (Active Comparator): Endurance training program of deep cervical flexors and deep cervical extensors with the conventional protocol.
  Interventions: Other: Conventional training protocol

INTERVENTIONS:
Other: Training protocol with the cervical device for treatment (CDAT). — Endurance training program of deep cervical flexors and deep cervical extensors with the cervical device for treatment.
  Arms: Experimental: Training protocol with the cervical device for treatment (CDAT).
Other: Conventional training protocol — Endurance training program of deep cervical flexors and deep cervical extensors with the conventional protocol.
  Arms: Conventional training protocol

SUMMARY:
The purpose of this study is to evaluate the clinical results in cervical spine range of motion, endurance deep cervical muscles, headache impact and physical activity enjoyment by a training protocol with the new device for cervical treatment (CDAT) versus conventional training protocol (CT) in subjects with cervicogenic headache.

DETAILED DESCRIPTION:
The cervical spine is the most mobile region of the spine and must be strong enough to support the weight of the skull. Strength deficits of the deep cervical muscles are related to different clinical conditions, such as cervicogenic headache. Cervicogenic headache is a secondary headache defined as a unilateral headache associated with neck pain, related to a decreased cervical range of motion and strength deficits of the deep cervical muscles.

Training protocols can help to improve pain, function, posture and cross-sectional area. However, there are no training protocols in subjects with cervicogenic headache including deep neck extensor and flexor muscles. The cervical device treatment (CDAT) allows us to train the cervical flexor and extensor muscle in a simple and comfortable way.

ELIGIBILITY:
Inclusion Criteria:

* Deep flexor strength deficit in craniocervical flexion test.
* Deep extensor strength deficit in neck extensor muscle endurance.
* A positive result in the flexion-rotation test
* ≥ 50 score in Headache Impact Test (HIT-6).
* Diagnosis of cervicogenic headache according to Sjaastad et al. Subjects will have to fulfill both parts I and III of the major criteria for diagnosis (pain aggravated by neck movement, sustained position or external pressure, restricted cervical range of motion, and unilateral pain starting in the neck and radiating to the frontotemporal region)

Exclusion Criteria:

* Have received head/cervical treatment during the last six month, presented any red flag, neurological or cognitive impairment (inability to understand the questionnaires or examination).
* Have received cervical manual therapy treatment during the last six month
* A history of head/cervical trauma or surgery during the last year.
* The use of pacemakers (the magnets in the CROM device could alter their signal
* Inability to perform the flexion-rotation test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2022-08-05 (Actual); Primary Completion 2022-10-15 (Actual); Study Completion 2022-11-15 (Actual)

PRIMARY OUTCOMES:
Change in Flexion Rotation Test (FRT) | Change between baseline and post intervention (6 weeks) and after 10 weeks.
  Mean change from baseline in Flexion-rotation test after 6 weeks and 10 weeks.
  The examiners assess the cervical ROM using CROM (Cervical Range-of-Motion Instrument). Flexion rotation test will be evaluated. Flexion rotation test is used to see the amount of movement of the upper cervical spine and is the test most used in the literature. It is positive when there is a decrease of 10 degrees or more in the cervical rotation with maximum flexion, in a sense with respect to the contralateral or presents hypomobility of segment C1 with a mobility less than 32.
Change in Headache Impact Test (HIT-6) (Headache Disfunction) | Change between baseline and post intervention (6 weeks) and after 10 weeks.
  Mean change from baseline in Headache Impact Test (HIT-6) after 6 weeks and 10 weeks.
  The examiners assess the impact of headache on patients' lives using the HIT-6. Very severe impact: 60 or more. Major impact: 56-59 score Some impact: 50-55 score Little or no impact: 49 or less.

SECONDARY OUTCOMES:
Craniocervical flexion test | Baseline and 6 weeks, 10 weeks.
  The examiners assess the strength of deep cervical flexors with craniocervical flexion test.
Cervical Spine Range of Motion (ROM). | Baseline and 6 weeks, 10 weeks.
  Mean change from baseline in Cervical Spine Range of Movement (ROM) after 6 weeks and 10 weeks.
  The examiners assess the cervical ROM using CROM (Cervical Range-of-Motion Instrument). Cervical flexion, extension, right/left sidebending, right/left rotation will be evaluated.
  The examiners assess the cervical ROM using CROM (Cervical Range-of-Motion Instrument). Upper cervical flexion, upper cervical extension will be evaluated.[Time Frame: Baseline and 6 weeks, 10 weeks]
Deep neck flexor endurance Test. | Baseline and 6 weeks, 10 weeks.
  Chin Tuck Neck Flexion Test is an assessment technique intended to determine the endurance of the deep cervical flexors.
Physical activity enjoyment Scale (PACES) | 6 weeks
  The examiners assess participant satisfaction with cervical deep muscle training.
  This scale measures enjoyment during physical activity through 16 items, which are preceded by the phrase "When I am active…" This instrument measures enjoyment and bipolar enjoyment, through statements such as "I enjoy it", "I'm bored", "It's very exciting", and "I don't like it". The answers will be collected on a Likert scale from 1 (totally disagree) to 5 (totally agree).

CONTACTS AND LOCATIONS:
Overall Officials: Pilar Pardos-Aguilella, Principal Investigator — UicCatalunya
Locations (1):
- Élite Fisioterapia, María Montessori 2., Zaragoza, Spain